CLINICAL TRIAL: NCT02299141
Title: A Pilot Study of Nintedanib in Molecularly Selected Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Nintedanib in Molecularly Selected Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201412116
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nintedanib (Experimental): -Nintedanib will be administered orally at a dose of 200 mg twice daily during each 28 day cycle. Starting with cycle 64, cycles will last 12 weeks.
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib
  Other Names: Ofev; BIBF 1120; Vargatef

SUMMARY:
There has been limited benefit with angiogenesis inhibitor drugs in molecularly unselected patients in non-small cell lung cancer (NSCLC). The investigators propose that patients who are molecularly selected for treatment with nintedanib based on the presence of mutations in the following genes: VEGFR1-3, PDGFR-A, PDGFR-B, FGFR1-3, and TP53, will have clinically meaningful benefit in terms of response rate (RR) and progression-free survival (PFS). Furthermore the investigators plan to correlate outcomes with specific mutations and evaluate mechanisms of resistance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced (metastatic or unresectable) NSCLC with mutations, rearrangement and fusion involving RET oncogene, or abnormalities (non-synonymous SNV or amplification) in the nintedanib target genes VEGFR1-3, TP53, PDGFR-A, PDGFR-B, and FGFR1-3. CLIA certified lab testing for nintedanib target genes using cell free DNA from peripheral blood and/or assays performed on tumor tissues are acceptable.
* Patients with EGFR mutations or ALK rearrangements must have disease progression on appropriate FDA-approved therapy for these genomic aberrations prior to enrollment.
* Disease progression on platinum-doublet chemotherapy prior to enrollment.
* At least one measurable lesion or evaluable disease. Measurable disease is defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm with CT scan, as ≥20 mm by chest x-ray, or ≥10 mm with calipers by clinical exam.
* Prior treatment of cancer (chemotherapy, radiation therapy, and surgery) is allowed if completed at least 3 weeks prior to start of treatment with nintedanib and if all treatment-related toxicities are resolved.
* At least 18 years of age.
* ECOG performance status 0-1
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9.0 g/dL
  * INR < 2.0
  * PT and PTT < 50% of deviation from IULN
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 1.5 x IULN for patients without liver metastases and ≤ 2.5 x IULN for patients with liver metastases
  * Urine protein < 2+
  * Creatinine within normal institutional limits OR Creatinine clearance > 45 mL/min for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 3 months after the end of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior treatment with VEGFR tyrosine kinase inhibitors.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Currently receiving any other investigational agents, or received an investigational agent within 3 weeks of the first dose of nintedanib.
* Radiotherapy to the target lesion within the past 3 months prior to baseline imaging.
* Symptomatic brain metastases. Patients with known brain metastases are eligible if the metastases are asymptomatic and previously treated.
* Leptomeningeal disease.
* Radiographic evidence of cavitary or necrotic tumors.
* Centrally located tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to nintedanib or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure > NYHA II, active coronary artery disease, unstable angina pectoris, serious cardiac arrhythmia, uncontrolled hypertension (defined as systolic pressures > 150 mmHg or diastolic pressure > 90 mmHg), pericardial effusion, uncontrolled seizure disorder, or psychiatric illness/social situations that would limit compliance with study requirements.
* Major injuries and/or surgery with then past 4 weeks prior to the start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period.
* History of clinically significant hemorrhagic or thromboembolic event in the past 6 months.
* Known inherited predisposition to bleeding or thrombosis.
* History of cardiac infarction within the past 12 months prior to the start of study treatment.
* Receiving therapeutic anticoagulation (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous device) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid < 325 mg QD).
* Pregnant and/or breastfeeding. Patients of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Significant weight loss (> 10% of BW) within past 6 months prior to inclusion into the trial.
* Known active or chronic hepatitis B or C infection.
* Active alcohol or drug abuse.
* Gastrointestinal disorder or abnormality that would interfere with absorption of the study drug.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with nintedanib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2025-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waqar SN, Rawat U, Morgensztern D, et al.; A pilot study of nintedanib in molecularly selected patients with advanced non-small cell lung cancer (NSCLC) (NCT02299141). J. Clin. Oncol. 38:15_suppl, e21694-e21694; (2020) URL: https://ascopubs.org/doi/abs/10.1200/JCO.2020.38.15_suppl.e21694
- [Derived] Auberle C, Gao F, Sloan M, Morgensztern D, Winkler L, Ward JP, Devarakonda S, Rearden TP, Govindan R, Waqar SN. A pilot study of nintedanib in molecularly selected patients with advanced non-small cell lung cancer. J Thorac Dis. 2024 Jun 30;16(6):3782-3793. doi: 10.21037/jtd-23-1717. Epub 2024 Jun 12. PMID 38983151
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Nintedanib: -Nintedanib will be administered orally at a dose of 200 mg twice daily during each 28 day cycle
Period: Overall Study
Arm/Group | Nintedanib
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nintedanib
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 66 [47 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: * RR = Partial response plus complete response using RECIST 1.1
  * Complete response (CR) = disappearance of all target lesions, non-target lesions, and normalization of tumor marker level
  * Partial response (PR) = at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline of sum diameters
Time Frame: After 2 cycles of therapy (approximately Day 56)
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib
Number analyzed (Participants) | 20
Participants | 3

2. Secondary Outcome: Median Progression-free Survival (PFS)
Description: * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease (PD) = at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, appearance of one or more non-target lesion(s) and/or unequivocal progression of existing non-target lesions
Time Frame: 12 months follow-up minimum
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nintedanib
Number analyzed (Participants) | 20
months | 4.3 [1.8 to 7.9]

3. Secondary Outcome: Response Rate by Mutation Type
Time Frame: At the time of response (approximately day 56)
Population: Only 3 participants had a response to treatment and are evaluable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib
Number analyzed (Participants) | 3
Participants
  TP53 mutation | 3
  PDGFR-A mutation | 0
  PDGFR-B mutation | 0
  FGFR1-3 mutation | 1
  VEGFR1-3 mutation | 0
  RET alteration | 0

4. Secondary Outcome: Unique Genetic Variations Associated With Extreme Responders (Both Non-responders and Responders)
Description: Correlate baseline genetic mutations with treatment response and progression of disease
Time Frame: Baseline and at the time of response (approximately Day 56)
Population: Only 7 participants are evaluable for this outcome measure as they were considered extreme responders.
Measure: Number; unit: mutations
Groups:
- Responder A: -Includes the mutations associated with Responder A
- Responder B: -Includes the mutations associated with Responder B
- Responder C: -Includes the mutations associated with Responder C
- Progressive Disease A: -Includes the mutations associated with participant Progressive Disease A
- Progressive Disease B: -Includes the mutations associated with participant Progressive Disease B
- Progressive Disease C: -Includes the mutations associated with participant Progressive Disease C
- Progressive Disease D: -Includes the mutations associated with participant Progressive Disease D
Arm/Group | Responder A | Responder B | Responder C | Progressive Disease A | Progressive Disease B | Progressive Disease C | Progressive Disease D
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
mutations
  TP53 C242F | 1 | 0 | 0 | 0 | 0 | 0 | 0
  TP53 A159V | 0 | 1 | 0 | 0 | 0 | 0 | 0
  TP53 A27V | 0 | 1 | 0 | 0 | 0 | 0 | 0
  TP53 P72R | 0 | 1 | 0 | 0 | 0 | 0 | 0
  TP53 M160_A161del | 0 | 0 | 1 | 0 | 0 | 0 | 0
  TP53 D281E | 0 | 0 | 0 | 1 | 0 | 0 | 0
  TP53 R342P | 0 | 0 | 0 | 0 | 1 | 0 | 0
  TP53 D207fs | 0 | 0 | 0 | 0 | 1 | 0 | 0
  TP53 Tyr234* | 0 | 0 | 0 | 0 | 0 | 1 | 0
  FGFR3 S249C | 1 | 0 | 0 | 0 | 0 | 0 | 0
  FGFR1 amplification | 0 | 0 | 0 | 0 | 0 | 0 | 1
  PDGFRA G166E | 0 | 0 | 0 | 1 | 0 | 0 | 0

5. Secondary Outcome: Genetic Mechanisms of Secondary Resistance
Description: Genomic analysis at time of progression after treatment with nintedanib (after response (complete response/partial response/stable disease) lasting for 6 months or longer) will provide some unique insights into mechanisms underlying acquired resistance.
Time Frame: At the time of progression (estimated to be 8 months)
Population: -Samples are available for 2 patients (1 patient with stable disease and 1 with partial response) but sample quantity not sufficient for genomic analysis.
Arm/Group | Nintedanib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: -Adverse events are collected from start of treatment until 30 days following the last day of study treatment.
Description: Only grade 3, 4, or 5 adverse events were collected per protocol unless a grade 1 or grade 2 event met the definition of an serious adverse event.
Arm/Group | Nintedanib
All-Cause Mortality (participants affected / at risk) | 12/20
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=20)
Atrial fibrillation (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Lung infection (Infections and infestations) | 3
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Confusion (Nervous system disorders) | 1
Edema cerebral (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Stroke (Nervous system disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=20)
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Drug induced liver injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT02299141/Prot_SAP_001.pdf